CLINICAL TRIAL: NCT01772277
Title: Efficacy of Mitomycin C in Endoscopic Dacryocystorhinostomy: A Systematic Review and Meta-Analysis
Status: Completed | Type: Observational
Sponsor: Yifan Feng (Other)
Collaborators: Wenzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Yifan Feng, Eye Hospital, Wenzhou Medical College, China, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: F20130115
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Dacryocystitis
Keywords: Endoscopic dacryocystorhinostomy; Mitomycin C
MeSH Terms: conditions — Dacryocystitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MMC group: patients were scheduled to undergo Endoscopic dacryocystorhinostomy with intraoperative MMC
- Control group: patients were scheduled to undergo Endoscopic dacryocystorhinostomy without intraoperative MMC

SUMMARY:
To assess the efficacy and safety of local application of intraoperative mitomycin C (MMC) at osteotomy site in endoscopic dacryocystorhinostomy(EN-DCR).

DETAILED DESCRIPTION:
Mitomycin C (MMC) is an antineoplastic agent that inhibits the synthesis of DNA, cellular RNA, and protein by inhibiting the synthesis of collagen by fibroblasts. MMC was originally used as a systemic chemotherapeutic agent, it has been widely used in ophthalmic practice both intraoperatively and postoperatively for prevention of pterygium recurrence, enhancing the success rate of glaucoma filtration surgery. Recently, use of MMC has been described in lacrimal drainage surgery. It is postulated that adjunctive use of MMC over the osteotomy site in endoscopic dacryocystorhinostomy(EN-DCR)surgery could inhibit scarring and granulation tissue formation around the osteotomy site or common canaliculus and enhance the success of EN-DCR surgery.

Many controlled trials have investigated adjunctive MMC for primary or revision EN-DCR to augment the surgical success rate, but the results are not completely consistent. To the best of our knowledge, there was no meta-analysis on comparison of success rate of EN-DCR with MMC (MMC group) and endoscopic dacryocystorhinostomy without MMC (control group). Therefore, the aim of this study was to undertake systematic review and meta-analysis to evaluate the efficacy of intraoperative MMC application in EN-DCR surgery and help ophthalmologists to determine whether it is a useful adjuvant in EN-DCR surgery.

ELIGIBILITY:
Inclusion Criteria:

1. comparative studies;
2. adult patients (> 18 years) with NLDO undergoing primary or revision EN-DCR;
3. all studies included were required to provide the success rates of both MMC and control groups, and the followed up time was more than 6 months.

Exclusion Criteria:

1. studies which did not provide the success rates;
2. studies which included pediatric cases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were scheduled to undergo endoscopic dacryocystorhinostomy and randomized to with and without MMC
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
success rate | 6 months
  Success was determined by the presence of any one of the following: (1) patent lacrimal passage on syringing, (2) symptomatic improvement, and (3) endoscopic visualisation of fluorescein dye at the nasal opening of the anastomoses.

SECONDARY OUTCOMES:
ostium size | 12 months
  Change of ostium size at 3-, 6- and 12-month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Shiming Cheng, MD, Principal Investigator — Eye Hospital, Wenzhou Medical College, China
Locations (1):
- Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Cheng SM, Feng YF, Xu L, Li Y, Huang JH. Efficacy of mitomycin C in endoscopic dacryocystorhinostomy: a systematic review and meta-analysis. PLoS One. 2013 May 13;8(5):e62737. doi: 10.1371/journal.pone.0062737. Print 2013. PMID 23675423